CLINICAL TRIAL: NCT00840151
Title: A SMART Design for Attendance-based Prize CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 09-053-2; P50DA009241-16 (NIH)
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Substance Abuse
Keywords: Substance Abuse; Contingency Management
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Group A (No Intervention): Individuals randomized to Treatment Group A will receive standard treatment for study weeks 1-6.
- Treatment Group B (Experimental): Individuals randomized to Treatment Group B will receive contingency management plus standard treatment for study weeks 1-6.
  Interventions: Behavioral: contingency management
- Aftercare Group A (No Intervention): All participants will be re-randomized after study week 6. Those participants assigned to Aftercare Group A will receive standard treatment for study weeks 7-12.
- Aftercare Group B (Experimental): All participants will be re-randomized after study week 6. Those participants assigned to Aftercare Group B will receive contingency management treatment plus standard treatment for weeks 7-12.
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Participants randomized to a contingency management treatment condition can earn the chance to win prizes for attending substance abuse treatment.
  Arms: Aftercare Group B; Treatment Group B

SUMMARY:
The purpose of this study is to compare different forms of treatment for substance abuse. This study will involve a type of treatment called contingency management, in which patients receive incentives (prizes) for attending outpatient treatment. This study will compare contingency management to standard treatment that does not involve incentives. This study will also compare contingency management treatment that lasts 6 weeks to contingency management that lasts 12 weeks. Finally, this study will compare contingency management treatment delivered at the beginning of outpatient treatment to contingency management treatment delivered later during outpatient treatment. The investigators hypothesize that (1) a 12-week attendance-based contingency management intervention will improve retention and enhance drug abstinence versus standard treatment, (2) initial short-term exposure to attendance-based contingency management (in weeks 1-6 only) will improve substance abuse treatment outcomes compared to standard treatment alone, and (3) contingency management in weeks 7-12 will be particularly useful for those with sporadic attendance or continued drug use during initial stages of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* current DSM-IV diagnosis of cocaine abuse or dependence or recent cocaine use (self-reported use in past 30 days or positive urine toxicology screen)
* willing to sign informed consent and able to pass an informed consent quiz

Exclusion Criteria:

* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk) on the basis of history or medical examination
* in recovery from pathological gambling (meet DSM-IV criteria for lifetime pathological gambling and are actively trying to refrain from gambling)
* do not speak English (all treatment is provided in English at these clinics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2009-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
longest duration of negative drug and alcohol samples submitted | throughout active phase and at each follow-up assessment

SECONDARY OUTCOMES:
proportions of samples testing negative for drugs and alcohol | during active phase and at each follow-up assessment
psychosocial functioning and HIV risk behaviors | baseline, active phase and at each follow-up assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States